CLINICAL TRIAL: NCT06462898
Title: Evaluate the Use of Omega-3 Fortified Smoothies to Improve Omega-3 Index and Physical Performance Related Outcomes Among Soldiers
Brief Title: The Effect of Omega-3 Fortified Smoothies on Omega-3 Index and Physical Performance Related Outcomes Among Soldiers
Acronym: H2FO3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Principal Investigator, Melissa Rittenhouse, Nutritionist/Exercise Scientist, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USUHS.2023-118
Record Dates: First submitted 2024-05-06; First posted 2024-06-17 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Nutrition, Healthy
Keywords: Omega-3 fatty acids; Holistic Health and Fitness (H2F); Army Combat Fitness Test (ACFT); Performance; Nutrition; Recovery

STUDY DESIGN:
Intervention Model Description: A blinded randomized-placebo control trial will be conducted in collaboration with the Army Holistic Health and Fitness (H2F) Program. Participants will be randomly selected from two H2F training sites: Ft. Campbell and Ft. Drum. In total, 100 participants will be randomly selected. Each site will have participants assigned to the placebo group and omega-3 enhanced smoothie group. Participants will be excluded if they have a fish allergy or if they are unable to complete an Army Combat Fitness Test (ACFT) for any reason. Participants taking omega-3 supplements will not be excluded, but will be instructed to be consistent for the duration of the study.
Who Masked: Participant
Masking Description: Participants will be blinded. The research team will pre-mix the drinks and have them labeled for participants daily. Both drinks look and taste the same.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omega-3 Fortified Protein Smoothie (Active Comparator): Participants will receive a shaker bottle containing 1 tbsp omega-3 powder and 1 scoop protein powder mixed with water, after morning physical training, five days a week, for eight weeks.
  Interventions: Dietary Supplement: Omega-3 Fortified Protein Smoothie
- Non-Fortified Protein Smoothie (Placebo Comparator): Participants will receive a shaker bottle containing 1 scoop protein mixed with water, after morning physical training, five days a week, for eight weeks.
  Interventions: Dietary Supplement: Non-Fortified Protein Smoothie

INTERVENTIONS:
Dietary Supplement: Omega-3 Fortified Protein Smoothie — Omega-3 powder and protein supplementation.
  Arms: Omega-3 Fortified Protein Smoothie
Dietary Supplement: Non-Fortified Protein Smoothie — Protein without omega-3 powder supplementation.
  Arms: Non-Fortified Protein Smoothie

SUMMARY:
The goal of this clinical trial is to test the effect of omega-3 on physical performance and recovery of Soldiers.

Objectives 1: Assess the impact of 8-weeks of daily consumption of 1600mg of omega-3 fortified smoothie on O3I response.

Objective 2: Determine the relationship between O3I and measures of performance and recovery.

Participants will:

* Be randomly assigned to placebo group or to the omega-3 fortified smoothie group.
* The intervention group will take omega-3 fortified smoothies and controls will consume a non-fortified smoothie, five days a week for 8 weeks.
* Participate in Army Combat Fitness Tests (ACFT)
* Complete surveys that assess dietary intake, physical activity (PAQ) and sleep quality (PSQI).
* Complete a finger prick to determine omega-3 index.

Assessments will be collected pre/post intervention. Researchers will compare intervention and placebo groups to see if omega-3 levels increase, and improve physical performance and recovery.

DETAILED DESCRIPTION:
Evidence suggests that mental and physical health are positively related to the omega-3 intake, and studies indicate that supplementation of omega-3 fatty acids may improve muscle recovery and range of motion while decreasing soreness and pain.

Omega-3 fatty acids are an essential part of the diet and are found primarily in marine-based sources of fatty fish including salmon, mackerel, and herring. The Omega-3 Index (O3I) is a reliable method used to measure omega-3 status, more specifically it represents the sum of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), as a percentage of red blood cells. Currently, O3I is the preferred method for assessing omega-3 status given its low biological variability and its ability to be measured in either the fed or fasted state. Generally, the O3I increases with greater consumption of marine-based omega-3; however, the extent varies by individual. Research indicates the general population and Service members alike have a low O3I (~4%) and therefore at risk for poor health and suboptimal physical performance. For optimal health, performance and a decreased risk for cardiovascular disease an O3I of ≥ 8 % is desirable.

The research utilizing the Omega-3 Index as a measure of omega-3 fatty acids began in relation to preventing severe cardiovascular risks. The research has expanded shows that omega-3 fatty acids can reduce triglyceride levels and may serve as an effective treatment option for cardiovascular disease, osteoporosis, psoriasis, and arthritis. Omega-3 fatty acids are thought to inhibit eicosanoids and inflammatory cytokines leading to analgesic effects. Additionally, preliminary studies support a rehabilitative role of omega-3 fatty acids in maintaining muscle mass and minimizing muscle wasting during a prolonged period of limb immobilization (i.e., leg cast). Furthermore, O3I levels have been positively correlated with muscle protein synthesis and enhanced recovery from muscle damaging exercise (i.e. delayed onset muscle soreness), in both athletic and military populations.

Improving Service Members health and maintaining the ability to perform optimally are high priorities. An average O3I of ~4% is concerning. These findings, although not surprising given the lack of foods containing omega-3 fatty acids across military installations, require action. Innovative solutions to provide Service Members with omega-3 fatty acids are needed to achieve health and performance benefits. Therefore, the purpose of this study is to examine whether increasing omega-3 fatty acid intake using a novel fortified food product improves performance and recovery outcomes in Holistic Health and Fitness (H2F) soldiers.

Researchers hypothesize regular consumption (one smoothie per day, five days per week, for eight weeks) of omega-3 fortified smoothies (1600 mg omega-3 per smoothie) will increase O3I to 8% compared to a control group. Researchers also hypothesize improvements in performance markers related to strength, flexibility, aerobic capacity and power as assessed by the Army Combat Fitness Test (ACFT), rate of perceived exertion (RPE), and recovery (a visual analog scale (VAS) for pain) in the intervention group compared to control. Researchers hypothesize the control group will not reach an O3I of 8% and measures of performance and recovery will be statistically lower than in the intervention group.

A blinded randomized-placebo control trial will be conducted in collaboration with the Army Holistic Health and Fitness (H2F) Program. Participants will be randomly selected from two H2F training sites: Ft. Campbell and Ft. Drum. In total, 100 participants will be randomly selected. Each site will have participants assigned to the placebo group and omega-3 enhanced smoothie group. Participants will be excluded if they have a fish allergy or if they are unable to complete an Army Combat Fitness Test (ACFT) for any reason. Participants taking omega-3 supplements will not be excluded, but will be instructed to be consistent for the duration of the study.

Previous research already indicates omega-3 status is low in military personal. Increasing omega-3 fatty acid intake will not only help maintain a healthy force by minimizing chronic disease risks, if researchers determine omega-3 fatty acids improve performance or recovery, guidelines can be developed and soldiers can be educated, possibly increasing the demand for these types of foods or alternatives will lead the way in improving the military nutrition environment.

ELIGIBILITY:
Inclusion Criteria:

* Active Duty Military Personnel
* Current soldier at Ft. Drum or Ft. Campbell.
* Able and willing to complete two Army Combat Fitness Test (ACFT) (Week 1 and week 8)
* Willing to obtain two finger pricks for the Omega-3 Index (week 1 and week 8)

Exclusion Criteria:

* Allergic to fish

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Omega-3 Index | Week 1 and Week 8
  Omega-3 Index will be measured through finger prick, obtaining 1-2 drops of blood on a collection card to be sent to OmegaQuant for analysis. A score of 8-12% is desirable, 4-7.9% is moderate and < 4% is low.
Army Combat Fitness Test (ACFT) | Week 1 and Week 8
  ACFT test will be performed at Week 1 baseline and Week 8 post-intervention to show changes in physical performance.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Rittenhouse, PhD, Principal Investigator — Uniformed Services University Health Sciences/Henry M. Jackson Foundation
Locations (2):
- United States (2):
  - Fort Campbell, Fort Campbell North, Kentucky
  - Fort Drum, Fort Drum, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Practice guideline for the treatment of patients with major depressive disorder (revision). American Psychiatric Association. Am J Psychiatry. 2000 Apr;157(4 Suppl):1-45. No abstract available. PMID 10767867
- [Background] Bozzatello P, De Rosa ML, Rocca P, Bellino S. Effects of Omega 3 Fatty Acids on Main Dimensions of Psychopathology. Int J Mol Sci. 2020 Aug 21;21(17):6042. doi: 10.3390/ijms21176042. PMID 32839416
- [Background] Colangelo LA, He K, Whooley MA, Daviglus ML, Liu K. Higher dietary intake of long-chain omega-3 polyunsaturated fatty acids is inversely associated with depressive symptoms in women. Nutrition. 2009 Oct;25(10):1011-9. doi: 10.1016/j.nut.2008.12.008. Epub 2009 Feb 4. PMID 19195841
- [Background] Guskiewicz KM, Marshall SW, Bailes J, McCrea M, Harding HP Jr, Matthews A, Mihalik JR, Cantu RC. Recurrent concussion and risk of depression in retired professional football players. Med Sci Sports Exerc. 2007 Jun;39(6):903-9. doi: 10.1249/mss.0b013e3180383da5. PMID 17545878
- [Background] Hibbeln JR. Fish consumption and major depression. Lancet. 1998 Apr 18;351(9110):1213. doi: 10.1016/S0140-6736(05)79168-6. No abstract available. PMID 9643729
- [Background] Hibbeln JR, Gow RV. The potential for military diets to reduce depression, suicide, and impulsive aggression: a review of current evidence for omega-3 and omega-6 fatty acids. Mil Med. 2014 Nov;179(11 Suppl):117-28. doi: 10.7205/MILMED-D-14-00153. PMID 25373095
- [Background] Johnston DT, Deuster PA, Harris WS, Macrae H, Dretsch MN. Red blood cell omega-3 fatty acid levels and neurocognitive performance in deployed U.S. Servicemembers. Nutr Neurosci. 2013 Jan;16(1):30-8. doi: 10.1179/1476830512Y.0000000025. Epub 2012 Jun 28. PMID 22748167
- [Background] Maes M, Smith R, Christophe A, Cosyns P, Desnyder R, Meltzer H. Fatty acid composition in major depression: decreased omega 3 fractions in cholesteryl esters and increased C20: 4 omega 6/C20:5 omega 3 ratio in cholesteryl esters and phospholipids. J Affect Disord. 1996 Apr 26;38(1):35-46. doi: 10.1016/0165-0327(95)00092-5. PMID 8735157
- [Background] Su KP, Matsuoka Y, Pae CU. Omega-3 Polyunsaturated Fatty Acids in Prevention of Mood and Anxiety Disorders. Clin Psychopharmacol Neurosci. 2015 Aug 31;13(2):129-37. doi: 10.9758/cpn.2015.13.2.129. PMID 26243838
- [Background] Teo L, Crawford C, Yehuda R, Jaghab D, Bingham JJ, Chittum HK, Gallon MD, O'Connell ML, Arzola SM, Berry K. Omega-3 polyunsaturated fatty acids to optimize cognitive function for military mission-readiness: a systematic review and recommendations for the field. Nutr Rev. 2017 Jun 1;75(suppl_2):36-48. doi: 10.1093/nutrit/nux008. PMID 28969342
- [Background] Weissman MM, Bland RC, Canino GJ, Faravelli C, Greenwald S, Hwu HG, Joyce PR, Karam EG, Lee CK, Lellouch J, Lepine JP, Newman SC, Rubio-Stipec M, Wells JE, Wickramaratne PJ, Wittchen H, Yeh EK. Cross-national epidemiology of major depression and bipolar disorder. JAMA. 1996 Jul 24-31;276(4):293-9. PMID 8656541
- [Background] Bucher HC, Hengstler P, Schindler C, Meier G. N-3 polyunsaturated fatty acids in coronary heart disease: a meta-analysis of randomized controlled trials. Am J Med. 2002 Mar;112(4):298-304. doi: 10.1016/s0002-9343(01)01114-7. PMID 11893369
- [Background] Patel A, Rova U, Christakopoulos P, Matsakas L. Assessment of Fatty Acids Profile and Omega-3 Polyunsaturated Fatty Acid Production by the Oleaginous Marine Thraustochytrid Aurantiochytrium sp. T66 Cultivated on Volatile Fatty Acids. Biomolecules. 2020 Apr 29;10(5):694. doi: 10.3390/biom10050694. PMID 32365742
- [Background] Gonzalez DE, McAllister MJ, Waldman HS, Ferrando AA, Joyce J, Barringer ND, Dawes JJ, Kieffer AJ, Harvey T, Kerksick CM, Stout JR, Ziegenfuss TN, Zapp A, Tartar JL, Heileson JL, VanDusseldorp TA, Kalman DS, Campbell BI, Antonio J, Kreider RB. International society of sports nutrition position stand: tactical athlete nutrition. J Int Soc Sports Nutr. 2022 Jun 23;19(1):267-315. doi: 10.1080/15502783.2022.2086017. eCollection 2022. PMID 35813846
- [Background] Kris-Etherton PM, Richter CK, Bowen KJ, Skulas-Ray AC, Jackson KH, Petersen KS, Harris WS. Recent Clinical Trials Shed New Light on the Cardiovascular Benefits of Omega-3 Fatty Acids. Methodist Debakey Cardiovasc J. 2019 Jul-Sep;15(3):171-178. doi: 10.14797/mdcj-15-3-171. PMID 31687095
- [Background] Rawson ES, Miles MP, Larson-Meyer DE. Dietary Supplements for Health, Adaptation, and Recovery in Athletes. Int J Sport Nutr Exerc Metab. 2018 Mar 1;28(2):188-199. doi: 10.1123/ijsnem.2017-0340. Epub 2018 Feb 19. PMID 29345167
- [Background] Vannice G, Rasmussen H. Position of the academy of nutrition and dietetics: dietary fatty acids for healthy adults. J Acad Nutr Diet. 2014 Jan;114(1):136-53. doi: 10.1016/j.jand.2013.11.001. PMID 24342605
- [Background] Black KE, Witard OC, Baker D, Healey P, Lewis V, Tavares F, Christensen S, Pease T, Smith B. Adding omega-3 fatty acids to a protein-based supplement during pre-season training results in reduced muscle soreness and the better maintenance of explosive power in professional Rugby Union players. Eur J Sport Sci. 2018 Nov;18(10):1357-1367. doi: 10.1080/17461391.2018.1491626. Epub 2018 Jul 9. PMID 29985775
- [Background] VanDusseldorp TA, Escobar KA, Johnson KE, Stratton MT, Moriarty T, Kerksick CM, Mangine GT, Holmes AJ, Lee M, Endito MR, Mermier CM. Impact of Varying Dosages of Fish Oil on Recovery and Soreness Following Eccentric Exercise. Nutrients. 2020 Jul 27;12(8):2246. doi: 10.3390/nu12082246. PMID 32727162
- [Background] Thielecke F, Blannin A. Omega-3 Fatty Acids for Sport Performance-Are They Equally Beneficial for Athletes and Amateurs? A Narrative Review. Nutrients. 2020 Nov 30;12(12):3712. doi: 10.3390/nu12123712. PMID 33266318
- [Background] Xin G, Eshaghi H. Effect of omega-3 fatty acids supplementation on indirect blood markers of exercise-induced muscle damage: Systematic review and meta-analysis of randomized controlled trials. Food Sci Nutr. 2021 Sep 21;9(11):6429-6442. doi: 10.1002/fsn3.2598. eCollection 2021 Nov. PMID 34760272
- [Background] Rittenhouse M, Scott J, Deuster P. Healthy Eating Index and Nutrition Biomarkers among Army Soldiers and Civilian Control Group Indicate an Intervention Is Necessary to Raise Omega-3 Index and Vitamin D and Improve Diet Quality. Nutrients. 2020 Dec 31;13(1):122. doi: 10.3390/nu13010122. PMID 33396252
- [Background] Durrington PN, Bhatnagar D, Mackness MI, Morgan J, Julier K, Khan MA, France M. An omega-3 polyunsaturated fatty acid concentrate administered for one year decreased triglycerides in simvastatin treated patients with coronary heart disease and persisting hypertriglyceridaemia. Heart. 2001 May;85(5):544-8. doi: 10.1136/heart.85.5.544. PMID 11303007
- [Background] Lovegrove JA, Lovegrove SS, Lesauvage SV, Brady LM, Saini N, Minihane AM, Williams CM. Moderate fish-oil supplementation reverses low-platelet, long-chain n-3 polyunsaturated fatty acid status and reduces plasma triacylglycerol concentrations in British Indo-Asians. Am J Clin Nutr. 2004 Jun;79(6):974-82. doi: 10.1093/ajcn/79.6.974. PMID 15159226
- [Background] Yzebe D, Lievre M. Fish oils in the care of coronary heart disease patients: a meta-analysis of randomized controlled trials. Fundam Clin Pharmacol. 2004 Oct;18(5):581-92. doi: 10.1111/j.1472-8206.2004.00268.x. PMID 15482380
- [Background] Rousseau JH, Kleppinger A, Kenny AM. Self-reported dietary intake of omega-3 fatty acids and association with bone and lower extremity function. J Am Geriatr Soc. 2009 Oct;57(10):1781-8. doi: 10.1111/j.1532-5415.2008.01870.x. PMID 18759757
- [Background] Weiss LA, Barrett-Connor E, von Muhlen D. Ratio of n-6 to n-3 fatty acids and bone mineral density in older adults: the Rancho Bernardo Study. Am J Clin Nutr. 2005 Apr;81(4):934-8. doi: 10.1093/ajcn/81.4.934. PMID 15817874
- [Background] Mayser P, Mrowietz U, Arenberger P, Bartak P, Buchvald J, Christophers E, Jablonska S, Salmhofer W, Schill WB, Kramer HJ, Schlotzer E, Mayer K, Seeger W, Grimminger F. Omega-3 fatty acid-based lipid infusion in patients with chronic plaque psoriasis: results of a double-blind, randomized, placebo-controlled, multicenter trial. J Am Acad Dermatol. 1998 Apr;38(4):539-47. doi: 10.1016/s0190-9622(98)70114-8. PMID 9555791
- [Background] Berbert AA, Kondo CR, Almendra CL, Matsuo T, Dichi I. Supplementation of fish oil and olive oil in patients with rheumatoid arthritis. Nutrition. 2005 Feb;21(2):131-6. doi: 10.1016/j.nut.2004.03.023. PMID 15723739
- [Background] Goldberg RJ, Katz J. A meta-analysis of the analgesic effects of omega-3 polyunsaturated fatty acid supplementation for inflammatory joint pain. Pain. 2007 May;129(1-2):210-23. doi: 10.1016/j.pain.2007.01.020. Epub 2007 Mar 1. PMID 17335973
- [Background] Miles EA, Calder PC. Influence of marine n-3 polyunsaturated fatty acids on immune function and a systematic review of their effects on clinical outcomes in rheumatoid arthritis. Br J Nutr. 2012 Jun;107 Suppl 2:S171-84. doi: 10.1017/S0007114512001560. PMID 22591891
- [Background] Edefonti V, Parpinel M, Ferraroni M, Boracchi P, Schioppo T, Scotti I, Ubiali T, Currenti W, De Lucia O, Cutolo M, Caporali R, Ingegnoli F. A Posteriori Dietary Patterns and Rheumatoid Arthritis Disease Activity: A Beneficial Role of Vegetable and Animal Unsaturated Fatty Acids. Nutrients. 2020 Dec 17;12(12):3856. doi: 10.3390/nu12123856. PMID 33348651
- [Background] McGlory C, Gorissen SHM, Kamal M, Bahniwal R, Hector AJ, Baker SK, Chabowski A, Phillips SM. Omega-3 fatty acid supplementation attenuates skeletal muscle disuse atrophy during two weeks of unilateral leg immobilization in healthy young women. FASEB J. 2019 Mar;33(3):4586-4597. doi: 10.1096/fj.201801857RRR. Epub 2019 Jan 10. PMID 30629458

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT06462898/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT06462898/ICF_001.pdf